CLINICAL TRIAL: NCT05795075
Title: Computerized Modified Paramedian Approach Technique（CMPAT） Versus Conventional Midline Approach Technique（MAT） of Lumbar Puncture: A Randomized Control Trial
Brief Title: Randomized Control Trial Comparing CMPAT and MAT for Lumbar Puncture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ChiCTR2300067937
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-04

CONDITIONS: a Randomized Controlled Trial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The involvement of patients and the public was not or will not be included in the design, implementation, reporting or dissemination of the research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerized Modified Paramedian Approach Technique (Experimental): The L3-4 inter-laminar space will be selected as the target for puncture, and in the longitudinal direction, 1.0-1.5cm will be opened beside the upper edge of the spinous process (tip) of the lower vertebra as the entry point. The lumbar puncture needle will be inserted vertically along the axis of the anesthesia needle. The puncture path will be maintained completely perpendicular to the skin until the needle reached the PLTLF (posterior layer of the thoracolumbar fascia), where some resistance will be felt. The puncture direction is adjusted as needed. The tip of the needle will be tilted 20±10° in the sagittal direction and 15±5° inward such that the tip will point at the midpoint of the spinal canal. After the needle reaches the PLTLF, it will be further inserted 3-7 cm.
  Interventions: Procedure: Computerized Modified Paramedian Approach Technique
- Conventional Midline Approach Technique (Experimental): Puncture will be performed on the posterior median line near the midpoint of the L3-4 Space of spinous process. The lumbar puncture needle will be inserted vertically along the axis of the anesthesia needle, or the tip of the needle will be tilted 15° in the sagittal direction toward the head, so that the needle path is parallel to the space of spinous process.
  Interventions: Procedure: Conventional Midline Approach Technique

INTERVENTIONS:
Procedure: Computerized Modified Paramedian Approach Technique — Computerized Modified Paramedian Approach Technique ( CMPAT )
  Arms: Computerized Modified Paramedian Approach Technique
Procedure: Conventional Midline Approach Technique — Conventional Midline Approach Technique
  Arms: Conventional Midline Approach Technique

SUMMARY:
The lumbar puncture (LP) technique is a widely utilized method for diagnosis and treatment purposes. Recently, the paramedian approach technique (PAT) has garnered increasing interest due to its advantages over the midline approach technique (MAT), which has traditionally been used for LP in clinical practice . Utilizing digital virtual human and computer simulation techniques, a new path has been proposed for the computerized modified paramedian approach technique (CMPAT). As such, the objective of the present study is to present a randomized controlled trial (RCT) protocol to investigate and compare the effects of CMPAT versus MAT in patients requiring LP.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years. Indication for LP.（Diagnostic lumbar puncture：Cerebrospinal fluid composition analysis，Cerebrospinal fluid pressure measurement；Cerebrospinal fluid release or lumbar Contiuous drainage of fluid，Intrathecal injection of lumbar cistern, etc.） Informed consent. Sufficient knowledge of the Chinese language to complete forms and follow instructions independently.

Exclusion Criteria:

* Cerebral hernia or high Cerebrospinal fluid pressure that might lead to Cerebral hernia.

Treatment with oral anticoagulant or anti-small plate(3 days or less)or coagulation disorders, various factors leading to a higher risk of bleeding.

Local infection or skin breakdown. Previous surgery on Lumbar spine segments. Pregnancy or lactation Severe somatic or psychiatric illness.（Severe anxiety or depression, etc.） Failure to be followed up as needed or worries about the potential risks of the study.

Failure to provide written informed consent or follow the protocol requirements.

Expected survival time being less than 1 month. Plan to emigrate within 1 month. Other conditions that are unsuitable for clinical research.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of puncture attempts in case of successful LP | 1 day
LP success rate | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No